CLINICAL TRIAL: NCT07216287
Title: Enhancing Cardiovascular Health in Mothers and Children Through Home Visiting (Supplement)
Brief Title: Sleep Health in Pregnant Women in ENRICH
Status: Not yet recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202508143; UH3HL162970 (NIH)
Record Dates: First submitted 2025-10-02; First posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Pregnancy; Sleep

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention, observational cohort study

SUMMARY:
This proposal will study sleep health in pregnant women who are of low socioeconomic status (SES) and are participating in the NHLBI-funded UH3 grant: "Enhancing Cardiovascular (CV) Health in Mothers and Children Through Home Visiting (ENRICH)". Objective sleep health will be measured using an in-home sleep disordered breathing testing device and actigraphy and associations of sleep health with social determinants of health and CV health will be investigated. Data from this study will serve as the foundation for future work that will result in the development of sleep interventions and updated guidelines for screening and treatment of sleep in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in a HV agency participating in ENRICH
2. Pregnant, with a single or multiple pregnancy, at or less than 34 weeks 0 days gestation
3. 18 years of age or older
4. low SES (Medicaid eligibility or income at or below the federal poverty line) and/or African American Race and/or Hispanic/Latino ethnicity

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A subset of 50 participants from the Washington University clinical center of ENRICH will be enrolled in this study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sleep Health | Baseline
  A sleep health index will be calculated using 7-day wrist actigraphy, a single overnight home SDB testing device, and questionnaires. A sleep health index will be calculated using 10 sleep health components. Each component will be dichotomized with 0 indicating "poor" and 1 indicating "healthy". Scores will range from 0-10 with 0 being the poorest and 10 being completely healthy sleep, a score <7 will indicate "poor sleep health".

IPD SHARING:
Plan to Share IPD: Yes
Data (sleep health metrics, demographic and social determinants of health metrics) resulting from this research will be shared via the Washington University School of Medicine (WUSM) institutional data repository, Digital Commons Data@Becker.
Time Frame: The sharable data produced by this project will be made accessible in a timely manner and no later than at the time of publication or by the end of the funding period, whichever occurs earlier. The duration of data preservation and sharing will be governed by the retention policies of Digital Commons Data@Becker
Access Criteria: Data will be de-identified prior to sharing in digital Digital Commons Data@Becker and will be made available via controlled access to the approved users who sign the DUA (data use agreement) to ensure the requestor has a legitimate reason for access, agrees not to attempt re-identification, and not to redistribute data to unauthorized users.